CLINICAL TRIAL: NCT01099839
Title: A Phase I Study to Assess Drug-Drug Interaction Between ASP1941 and Miglitol.
Brief Title: A Study to Assess Drug-Drug Interaction Between ASP1941 and Miglitol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-0062
Record Dates: First submitted 2010-03-30; First posted 2010-04-08 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP1941
Keywords: ASP1941; Miglitol
MeSH Terms: interventions — ipragliflozin; miglitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one group (Experimental): Subjects will receive "ASP1941 alone", "Miglitol alone" and "ASP1941 + Miglitol" in different order.
  Interventions: Drug: ASP1941; Drug: Miglitol

INTERVENTIONS:
Drug: ASP1941 — oral
Drug: Miglitol — oral
  Other Names: Seibule

SUMMARY:
This study is to assess the pharmacokinetic interaction between ASP1941 and Miglitol in healthy volunteers.

DETAILED DESCRIPTION:
This will be a randomized, open-label, 3-way crossover design study to assess the drug-drug interaction between a single oral dose of ASP1941 and a single oral dose of Miglitol in healthy adult male volunteers. Each subject will receive "ASP1941 alone", "Miglitol alone" and "ASP1941 + Miglitol".

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and laboratory tests
* Body weight ; ≥50.0 kg, <80.0 kg
* Body Mass Index ; ≥17.6, <26.4
* Written informed consent has been obtained

Exclusion Criteria:

* Received any investigational drugs within 120 days before the screening assessment
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the screening assessment
* Received medication within 7 days before hospital admission
* A deviation from the assessment criteria of physical examinations or laboratory tests at screening or upon admission
* History of drug allergies
* With renal, hepatic, gastrointestinal, heart, cerebrovascular or respiratory diseases
* Previous treatment with ASP1941

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP1941 and Miglitol through analysis of blood samples | For 72 hours after each administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan